CLINICAL TRIAL: NCT01415245
Title: Vein External Support Trial
Acronym: VEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Graft Solutions Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CI-01-01
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Device applied to saphenous vein graft
  Interventions: Device: Fluent (VGS Fluent external support device)
- Control (No Intervention): Saphenous vein graft without device support

INTERVENTIONS:
Device: Fluent (VGS Fluent external support device) — Fluent external support device applied to saphenous vein graft
  Arms: Treatment

SUMMARY:
Prospective, multi-center, randomized, controlled pilot study to demonstrate the safety and effectiveness of the VGS Fluent external support device, supporting saphenous vein grafts in patients with coronary heart disease.

ELIGIBILITY:
Primary Inclusion Criteria:

1. Patient scheduled for on-pump CABG on clinical grounds
2. Vein grafts indicated for right and circumflex coronary arteries and LIMA indicated for the LAD on clinical grounds
3. Native circumflex and right coronary arteries have at least one stenosis in each vessel> 75%

Primary Exclusion Criteria:

1. Concomitant non-CABG cardiac procedure
2. Prior peripheral vascular or cardiac surgery
3. Emergency CABG surgery (cardiogenic shock, inotrophic pressure support, IABP)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Royal Brompton Hospital, London
  - Harefield Hospital, Middlesex
  - The John Radcliffe Hospital, Oxford

REFERENCES:
- [Derived] Taggart DP, Webb CM, Desouza A, Yadav R, Channon KM, De Robertis F, Di Mario C. Long-term performance of an external stent for saphenous vein grafts: the VEST IV trial. J Cardiothorac Surg. 2018 Nov 19;13(1):117. doi: 10.1186/s13019-018-0803-9. PMID 30453984